CLINICAL TRIAL: NCT02593851
Title: A Phase 1b, Randomized, Partially Double-blind, Placebo-controlled Study to Assess the Pharmacokinetics, Safety, and Tolerability of Multiple Doses of Orally Administered JNJ-53718678 in Infants Hospitalized With RSV Infection
Brief Title: A Study to Assess the Pharmacokinetics, Safety, and Tolerability of Multiple Doses of Orally Administered JNJ-53718678 in Infants Hospitalized With Respiratory Syncytial Virus (RSV) Infection
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Trial was cancelled due to availability of clinical supplies.
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR107945; 2015-002003-28 (EudraCT Number); 53718678RSV1005 (Other: Janssen Sciences Ireland UC)
Record Dates: First submitted 2015-08-21; First posted 2015-11-02 (Estimated); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Respiratory Syncytial Virus Infections; Virus Diseases
Keywords: Respiratory Syncytial Virus Infections; JNJ-53718678; Placebo; Infants
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Virus Diseases | interventions — JNJ-53718678

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (16):
- Part 1: Cohort 1a (Experimental): Participants (greater than or equal to [>=] 6 months and less than or equal to [<=] 24 months of age) will receive JNJ-53718678, 2 milligram per kilogram body weight (mg/kg) oral solution once daily on Day 1 to Day 7. Dose and/or dosing regimen may be adapted in subsequent cohorts based on the review of the safety/tolerability and full pharmacokinetic data from Cohort 1a.
  Interventions: Drug: JNJ-53718678
- Part 1: Cohort 1b (Experimental): Participants (>= 6 months and <= 24 months of age) will receive total daily dose of 6 mg/kg JNJ-53718678 oral solution or placebo [either in once daily [qd] or twice daily [bid]) on Day 1 to Day 7.
  Interventions: Drug: JNJ-53718678; Drug: Placebo
- Part 1: Cohort 1c (Experimental): Participants (>= 6 months and <= 24 months of age) will receive total daily dose of 18 mg/kg JNJ-53718678 oral solution or placebo [either in a qd or a bid regimen] on Day 1 to Day 7.
  Interventions: Drug: JNJ-53718678; Drug: Placebo
- Part 1: Cohort 1d (Experimental): Participants (>= 6 months and <= 24 months of age) will receive JNJ-53718678 oral solution or placebo [either in a qd or a bid regimen] on Day 1 to Day 7. The cohort 1d is optional and may be included at the discretion of the sponsor.
  Interventions: Drug: JNJ-53718678; Drug: Placebo
- Part 1: Cohort 1e (Experimental): Participants (>= 6 months and <= 24 months of age) will receive JNJ-53718678 oral solution or placebo [either in a qd or a bid regimen] on Day 1 to Day 7. The cohort 1e is optional and may be included at the discretion of the sponsor.
  Interventions: Drug: JNJ-53718678; Drug: Placebo
- Part 1: Cohort 2a (Experimental): Participants (>= 3 months and less than [<] 6 months of age) will receive total daily dose of 1.5 mg/kg JNJ-53718678 oral solution [either in a qd or a bid regimen] on Day 1 to Day 7.
  Interventions: Drug: JNJ-53718678
- Part 1: Cohort 2b (Experimental): Participants (>=3 months and < 6 months of age) will receive total daily dose of 4.5 mg/kg JNJ-53718678 oral solution or placebo [either in a qd or a bid regimen] on Day 1 to Day 7.
  Interventions: Drug: JNJ-53718678; Drug: Placebo
- Part 1: Cohort 2c (Experimental): Participants (>= 3 months and < 6 months of age) will receive total daily dose of 13.5 mg/kg JNJ-53718678 oral solution or placebo [either in a qd or a bid regimen] on Day 1 to Day 7
  Interventions: Drug: JNJ-53718678; Drug: Placebo
- Part 1: Cohort 2d (Experimental): Participants (>= 3 months and < 6 months of age) will receive JNJ-53718678 oral solution or placebo [either in a qd or a bid regimen] on Day 1 to Day 7. The cohort 2d is optional and may be included at the discretion of the sponsor.
  Interventions: Drug: JNJ-53718678; Drug: Placebo
- Part 1: Cohort 2e (Experimental): Participants (>= 3 months and < 6 months of age) will receive JNJ-53718678 oral solution or placebo [either in a qd or a bid regimen] on Day 1 to Day 7. The cohort 2e is optional and may be included at the discretion of the sponsor.
  Interventions: Drug: JNJ-53718678; Drug: Placebo
- Part 1: Cohort 3a (Experimental): Participants (greater than (>) 1 month and < 3 months of age) will receive total daily dose of 1 mg/kg JNJ-53718678 oral solution [either in a qd or a bid regimen] on Day 1 to Day 7.
  Interventions: Drug: JNJ-53718678
- Part 1: Cohort 3b (Experimental): Participants (> 1 month and < 3 months of age) will receive total daily dose of 3 mg/kg JNJ-53718678 oral solution or placebo [either in a qd or a bid regimen] on Day 1 to Day 7.
  Interventions: Drug: JNJ-53718678; Drug: Placebo
- Part 1: Cohort 3c (Experimental): Participants (> 1 month and < 3 months of age) will receive total daily dose of 9 mg/kg JNJ-53718678 oral solution or placebo [either in a qd or a bid regimen] on Day 1 to Day 7.
  Interventions: Drug: JNJ-53718678; Drug: Placebo
- Part 1: Cohort 3d (Experimental): Participants (> 1 month and < 3 months of age) will receive JNJ-53718678 oral solution or placebo [either in a qd or a bid regimen] on Day 1 to Day 7. The cohort 3d is optional and may be included at the discretion of the sponsor.
  Interventions: Drug: JNJ-53718678; Drug: Placebo
- Part 1: Cohort 3e (Experimental): Participants (> 1 month and < 3 months of age) will receive JNJ-53718678 oral solution or placebo [either in a qd or a bid regimen] on Day 1 to Day 7. The cohort 3e is optional and may be included at the discretion of the sponsor.
  Interventions: Drug: JNJ-53718678; Drug: Placebo
- Part 2: Cohort f (Experimental): Participants of all age groups will receive daily dose of JNJ-53718678 oral solution or placebo, either in a qd or a bid regimen on Days 1 to 7.
  Interventions: Drug: JNJ-53718678; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-53718678 — JNJ-53718678 oral solution will be administered once or twice daily for 7 days.
Drug: Placebo — Placebo oral solution will be administered once or twice daily for 7 days.
  Arms: Part 1: Cohort 1b; Part 1: Cohort 1c; Part 1: Cohort 1d; Part 1: Cohort 1e; Part 1: Cohort 2b; Part 1: Cohort 2c; Part 1: Cohort 2d; Part 1: Cohort 2e; Part 1: Cohort 3b; Part 1: Cohort 3c; Part 1: Cohort 3d; Part 1: Cohort 3e; Part 2: Cohort f

SUMMARY:
The purpose of this study is to evaluate pharmacokinetics, safety, tolerability, antiviral activity, and impact on the clinical course of Respiratory Syncytial Virus (RSV) infection after multiple oral doses of JNJ-53718678 at different doses and/or dosing regimens in infants (greater than [>] 1 month to less than or equal to [<=] 24 months of age) who are hospitalized with RSV infection.

DETAILED DESCRIPTION:
This is a Phase 1b, randomized (study medication assigned to participants by chance), partially double-blind (neither physician nor participant knows the identity of the assigned treatment), placebo-controlled, multicenter, multiple ascending dose study of JNJ 53718678 in infants (greater than [>] 1 month to less than or equal to [<=] 24 months of age) who are hospitalized with RSV infection. The duration of study will be approximately 4 weeks for each participant excluding screening period. In Part 1 of study, minimum total number of 42 participants will be divided in 3 cohorts: Age group 1 (Cohorts 1a-1e) (greater than or equal to [>=] 6 months and less than or equal to [<=] 24 months of age), Age group 2 (Cohorts 2a-2e)(>=3 months and less than [<] 6 months of age) and Age group 3 (Cohorts 3a-3e) (greater than [>] 1 month and <3 months of age). Each age group will consist of a minimum of 3 cohorts with the possibility to add 2 more per age group (Cohorts a through e) in which different doses and/or dosing regimens will be evaluated. Each cohort will consist of 5 participants (4 participants receiving JNJ-53718678 and 1 participant receiving placebo for 7 days), except for the first cohort of each age group which will contain only 4 participants (4 participants receiving JNJ 53718678). In Part 2 of the study, all age groups will be included in a single cohort, Cohort f, in which the selected dose regimen determined during Part 1 of the study will be used for each of the 3 age groups. A minimum of approximately 18 (12 participants receiving JNJ 53718678 and 6 participants receiving placebo) and a maximum of 24 participants (16 participants receiving JNJ 53718678 and 8 participants receiving placebo) will be included in this part of the study. Pharmacokinetics and safety of JNJ-53718678 will be evaluated primarily. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant has presented at the hospital for suspected Respiratory Syncytial Virus (RSV) infection within 72 hours prior to Screening completion
* Participant has been hospitalized for this suspected RSV infection
* Participant has been diagnosed with RSV infection using a polymerase chain reaction (PCR)-based assay, preferably commercially available locally
* Participant was born after a normal term pregnancy (greater than or equal to 37 weeks and 0 days)
* A legally acceptable representative of the participant must sign an Informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study, are willing for their child to participate in the study, are willing for their child to remain in the hospital for the first 3 days of dosing (even if not clinically indicated), and are willing/able to adhere to the prohibitions and restrictions specified in the protocol and study procedures

Exclusion Criteria:

* Participant who had major surgery within the 28 days prior to randomization or planned major surgery through the course of the study
* Participant has major congenital anomalies or known cytogenetic disorders
* Participant has known or suspected immunodeficiency, such as known human immunodeficiency virus (HIV) infection
* Participant has known or suspected hepatitis B or C infection
* Participant is upon current admission initially hospitalized in the Intensive care unit (ICU) and/or in need of invasive endotracheal mechanical ventilation

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2015-12-04 (Actual); Primary Completion 2017-03-21 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of JNJ-53718678 | Days 1, 2 and 3
  The Cmax is the maximum observed plasma concentration.
Trough Plasma Concentration (Ctrough) of JNJ-53718678 | Days 1, 2 and 3
  The Ctrough is the plasma concentration before dosing or at the end of the dosing interval of any dose other than the first dose in a multiple dosing regimen.
Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) | Days 1, 2 and 3
  The AUCtau is the measure of the plasma drug concentration from time zero to end of dosing interval.
Total Apparent Clearance (CL/F) of JNJ-53718678 | Days 1, 2 and 3
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vd/F) of JNJ-53718678 | Days 1, 2 and 3
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vd/F) is influenced by the fraction absorbed.
Number of Participants With Adverse Events | Up to Follow-up (Day 28)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

SECONDARY OUTCOMES:
Area Under the Viral Load-time Curve (VL AUC) | Up to Follow-up (Day 28)
  VL will be determined by quantitative real-time reverse transcriptase-polymerase chain reaction (qRT-PCR) assay of nasal swabs. The VL AUC (copies. hour/ml) will be calculated based on the trapezoidal method.
Amount of Viral Load Over Time | Up to Follow-up (Day 28)
  VL (copies/ml) at each assessment timepoint where a nasal sample is obtained.
Number of viral particles at Peak Viral Load | Up to Follow-up (Day 28)
  Peak viral load (copies/ml) is a measure of the maximum number of viral particles present in nasal swabs.
Time To Peak Viral Load | Up to Follow-up (Day 28)
  Time (hours) to peak viral load will be reported.
Number of Participants Reaching Undetectability of virus Between First Administration of Study Drug and Day 28 | Day 1 to Day 28
  Non-detectability of virus in nasal swabs between first administration of study drug and Day 28 will be reported.
Total Number of Respiratory Syncytial Virus (RSV) Hospitalization Days from Admission to Discharge | Up to Follow-up (Day 28)
  The total number of Respiratory Syncytial Virus (RSV) hospitalization days from admission to discharge will be reported.
Total RSV Hospitalization Days with Supplemental Oxygen Requirement | Up to Follow-up (Day 28)
  The total number of RSV Hospitalization Days with Supplemental Oxygen Requirement will be reported.
The Number of days in Intensive care unit (ICU) due to RSV | Up to Follow-up (Day 28)
  The number of days stayed in ICU due to RSV will be reported.
Total Days of non-invasive ventilator support During RSV Hospitalization | Up to Follow-up (Day 28)
  The total number of days with non-invasive ventilator support during RSV hospitalization will be reported.
Total Days of Mechanical Ventilation During RSV Hospitalization | Up to Follow-up (Day 28)
  The total number of days with Mechanical Ventilation during RSV hospitalization will be reported.
Changes in Peripheral Capillary Oxygen Saturation (SpO2) | Up to Follow-up (Day 28)
  The Percentage of Peripheral Capillary Oxygen Saturation (SpO2) will be assessed by the investigator during hospitalisation.
Change from Baseline in Respiratory Rate | Up to Follow-up (Day 28)
  The Respiratory rate (number of breaths per minute) will be assessed by the investigator and caregiver during hospitalisation.
Change from Baseline in Body Temperature | Up to Follow-up (Day 28)
  The body temperature (degrees Celcius) will be assessed by the investigator and caregiver during hospitalisation.
Clinical Symptom Score | Up to Follow-up (Day 28)
  The clinical symptom score will be assessed by the investigator (Clinician Outcome Assessment) and caregiver symptom Diary for each symptom. Clinical Symptom score ranges from 0 (best) to 4 (worst).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trial, Study Director — Janssen Sciences Ireland UC
Locations (39):
- Kirksville, Missouri, United States
- Argentina (3):
  - Bahía Blanca
  - City of Buenos Aires
  - Córdoba
- Australia (3):
  - Geelong
  - Hobart
  - Westmead
- Belgium (6):
  - Anderlecht
  - Brussels
  - Charleroi
  - Edegem
  - Leuven
  - Lier
- Brazil (5):
  - Curitiba
  - Porto Alegre
  - Ribeirão Preto
  - Rio de Janeiro
  - São Paulo
- Germany (4):
  - Freiburg im Breisgau
  - Hamm
  - Heidelberg
  - München
- Netherlands (2):
  - Hoofddorp
  - Utrecht
- Philippines (2):
  - Cebu City
  - Manila
- Spain (9):
  - Almería
  - Barcelona
  - Esplugues de Llobregat
  - Getafe
  - Madrid
  - Málaga
  - Santiago de Compostela
  - Seville
  - Valencia
- Sweden (4):
  - Gothenburg
  - Linköping
  - Lund
  - Malmo

REFERENCES:
- [Derived] Martinon-Torres F, Rusch S, Huntjens D, Remmerie B, Vingerhoets J, McFadyen K, Ferrero F, Baraldi E, Rojo P, Epalza C, Stevens M. Pharmacokinetics, Safety, and Antiviral Effects of Multiple Doses of the Respiratory Syncytial Virus (RSV) Fusion Protein Inhibitor, JNJ-53718678, in Infants Hospitalized With RSV Infection: A Randomized Phase 1b Study. Clin Infect Dis. 2020 Dec 17;71(10):e594-e603. doi: 10.1093/cid/ciaa283. PMID 32201897